CLINICAL TRIAL: NCT02981589
Title: Weaning Outcome From Invasive Mechanical Ventilation: a Prospective, Observational Cohort Study
Brief Title: Weaning Outcome From Invasive Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, MD, Beijing Chao Yang Hospital
Other Study IDs: BeijingCYH-ICU-003
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Patients Requiring Endotracheal Intubation and Invasive Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Invasive mechanical ventilation — Invasive ventilation was performed to all eligible patients. When patients met predefined criteria, spontaneous breathing trial was performed. Given spontaneous breathing trial passed, patients were extubated; on the contrary, patients would continue to receive invasive ventilation. If patients had respiratory failure after extubation, reintubation and invasive ventilation were necessary.

SUMMARY:
The main purpose of the present study was to explore the weaning failure rate from invasive mechanical ventilation and to identify risk factors of weaning failure.

ELIGIBILITY:
Inclusion Criteria:

* Requiring endotracheal intubation and invasive mechanical ventilation

Exclusion Criteria:

* Duration of invasive mechanical ventilation < 48 hours；
* Presence of tracheostomy；
* Presence of upper airway obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring endotracheal intubation and invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2023-12 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Weaning failure rate | 3.5 years
Spontaneous breathing trial failure rate | 3.5 years
Extubation failure rate | 3.5 years

SECONDARY OUTCOMES:
ICU mortality | 3.5 years
Hospital mortality | 3.5 years
ICU length of stay | 3.5 years
Hospital length of stay | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zujin Luo, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Respiratory intensive care unit, Beijing Chao Yang Hospital Jingxi Campus, Beiling, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Z, Zheng Y, Yang L, Liu S, Zhu J, Zhao N, Pang B, Cao Z, Ma Y. Neutrophil/lymphocyte ratio is helpful for predicting weaning failure: a prospective, observational cohort study. J Thorac Dis. 2018 Sep;10(9):5232-5245. doi: 10.21037/jtd.2018.08.68. PMID 30416770